CLINICAL TRIAL: NCT01881568
Title: Efficacy of Topical Tranexamic Acid Versus Intravenous Administration to Reduce Blood Transfusion Rate in Total Knee Arthroplasty Surgery: Phase III, Unicentric, Controlled,Double Blind, Randomized Non Inferiority Clinical Trial.
Brief Title: Efficacy Comparison of Topical and Intravenous Tranexamic Acid to Reduce the Number of Blood Transfusions in TKA
Acronym: TRANEX1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital Universitario La Paz (Other)
Responsible Party: Principal Investigator, Enrique Gómez Barrena, Professor, Hospital Universitario La Paz
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TRANEX1
Record Dates: First submitted 2013-02-05; First posted 2013-06-19 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Blood Loss
Keywords: Total Knee Arthroplasty, TKA, blood loss
MeSH Terms: conditions — Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental (Experimental): 1. Topical administration of 3g of Tranexamic Acid in 100mL of normal saline (0.9% sodium chloride) as follow:
     * 50mL by irrigation before wound closure
     * 50mL by intraarticular administration (Drenofast) after wound closure.
  2. Intravenous administration of Normal saline (0.9% sodium chloride) as follow:
     * 100mL before tourniquet realised
     * 100mL 3 hours after surgery
  Interventions: Drug: Tranexamic Acid
- Comparator (Active Comparator): 1. Topical administration of Normal saline (0.9% sodium chloride) as follow:
     * 50mL by irrigation before wound closure
     * 50mL by intraarticular administration (Drenofast) after wound closure
  2. Intravenous administration of two dosis of Tranexamic Acid as follow:
     * 15mg/kg of Tranexamic Acid in 100mL of normal saline (0.9% sodium chloride), before tourniquet realised
     * 15mg/kg of Tranexamic Acid in 100mL of normal saline (0.9% sodium chloride), 3 hours after surgery
  Interventions: Drug: Tranexamic Acid

INTERVENTIONS:
Drug: Tranexamic Acid — Topical administration: 3g of Tranexamic Acid in 100mL of normal saline (0.9% sodium chloride)
  Other Names: AMCHAFIBRIN
  Arms: Experimental
Drug: Tranexamic Acid — Intravenous administration of two dosis of Tranexamic Acid (15mg/kg of Tranexamic Acid in 100mL of normal saline each)
  Other Names: AMCHAFIBRIN,
  Arms: Comparator

SUMMARY:
The main objective is to evaluate the efficacy and safety of topical Tranexamic Acid (TA) to reduce the blood transfusion rate in total knee arthroplasty. The secondary endpoints are to estimate the visible blood loss at 24 hours after surgery, and invisible blood loss through serial counting of Hb/Htc. Methodology. TRANEX1 is a phase III, unicentric, controlled, randomized, double blind clinical trial that compare efficacy and safety of topical TA versus intravenous TA in a multimodal protocol, with no-inferiority criteria(n=79).

DETAILED DESCRIPTION:
The groups will be compared by ITT and PP. The non-inferiority would be estimated by comparing the confidence interval using the traditional test, and Wilson test.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (greater than 18 years old)
* Patients scheduled for primary unilateral knee arthroplasty
* Patients for La Paz- Cantoblanco Hospital, Madrid, Spain

Exclusion Criteria:

* Patients that refuse to sign the Inform Consent
* Allergy to tranexamic acid
* Major comorbidities: Severe ischemic heart disease(class III and IV of New York Heart Association); sleep apnea syndrome; severe EPOC; renal dysfunction (plasma creatinine>2mg/dL if mens and >1.8mg/dL if woman); or hepatic disfunction.
* Coagulopathy (preoperative platelet count <150,000/mm3, INR>1.4, prolonged PPT(>1.4 x normal)
* History of thromboembolic disease: CVA, DVT, PE
* Blood dyscrasias
* Retinopathy (disturbances of color vision)
* Jehovah's witnesses
* Pregnancy
* Breastfeeding
* Been participating or been participated a year ago in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2013-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Blood transfusion rate | participants will be followed for the duration of hospital stay, an expected average of 5 days
  Number of transfused patients in each arm/Total number of patients in each arm

SECONDARY OUTCOMES:
Visible blood loss | 24 hours after surgery
  Number of milliliters drained in Redon after 24 hours post OP
Invisible blood loss | 48 hours after surgery
  Number of milliliters estimated with Nedler formula 48 hours after surgery. Invisible blood loss= 75*weight(Kg)*[(Hb0-Hb1)/Hb0]+ blood transfused(mL)
Surgery infection rate | One month after surgery
  * Percent of patients with proved signs of infection during the hospital stay
  * Percent of patients with proved signs of infection one month after surgery(safety reasons)
Range of motion | participants will be followed for the duration of hospital stay, an expected average of 5 days
  - Range (in degrees) from full extension to full flexion during the hospital stay
Prevalence of drug-related adverse events | participants will be followed for the duration of hospital stay, an expected average of 5 days
  Rate and characteristics of the adverse events during the hospital stay
Rate of PE | One month after surgery
  * Percent of PE during the hospital stay
  * Percent of PE one month after surgery(safety reasons)
Rate of DVT | One month after surgery
  * Percent of DVT during the hospital stay
  * Percent of DVT one month after surgery(safety reasons)
Rate or Thrombophlebitis | One month after surgery
  * Percent of Thrombophlebitis during the hospital stay
  * Percent of Thrombophlebitis one month after surgery(safety reasons)

CONTACTS AND LOCATIONS:
Overall Officials: Enrique Gomez Barrena, PI, Principal Investigator — Hospital Universitario La Paz
Locations (1):
- Hospital Universitario La Paz, Madrid, Madrid, Spain

REFERENCES:
- [Derived] Gomez-Barrena E, Ortega-Andreu M, Padilla-Eguiluz NG, Perez-Chrzanowska H, Figueredo-Zalve R. Topical intra-articular compared with intravenous tranexamic acid to reduce blood loss in primary total knee replacement: a double-blind, randomized, controlled, noninferiority clinical trial. J Bone Joint Surg Am. 2014 Dec 3;96(23):1937-44. doi: 10.2106/JBJS.N.00060. PMID 25471907